CLINICAL TRIAL: NCT06652646
Title: MBOTE-Kamituga / Mpox Biology, Outcome, Transmission and Epidemiology - Protocole De Caractérisation Clinique Et Virologique Des Infections À Virus De Monkeypox À Kamituga (MBOTE-Kamituga)
Brief Title: Mpox Biology, Outcome, Transmission and Epidemiology
Status: Enrolling by invitation | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Ministry of Public Health, Democratic Republic of the Congo (Other Government); Research Foundation Flanders (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Project 427100 MPX
Record Dates: First submitted 2024-10-11; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Mpox (Monkeypox)
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 59 Days
Biospecimen Retention: Samples With DNA — skin swab, oropharyngeal swab, saliva, urine, semen, breast milk, anal swab, vaginal swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The MBOTE-Kamituga clinical and virological characterization protocol is a prospective observational cohort study with clinical and virological description of suspected mpox cases and longitudinal follow-up of confirmed mpox cases. Research activities will be aligned as far as possible with the response to the epidemic.

DETAILED DESCRIPTION:
For several decades, the Democratic Republic of Congo (DRC) has been the country most affected by monkeypox. While the global monkeypox epidemic (commonly known as mpox) of 2022-2023 was caused by clade II monkeypox virus (VMPX), outbreaks in the DRC are caused by the more virulent clade I variant. In recent years, and particularly in 2023, the country has seen a sharp increase in the number of cases, as well as a geographical expansion of the disease, with previously unaffected regions now reporting cases. Until recently, VMPX infections in the DRC were thought to be primarily the result of zoonotic transmission, with rather limited secondary human-to-human transmission. However, in recent months, an increasing number of cases linked to sexual transmission of clade I have been reported.

The Kamituga health zone is a densely populated mining region in South Kivu. The region reported no cases of smallpox in recent decades until, in October 2023, the disease was detected for the first time and began to affect mainly adolescents and young adults. To date, nearly 200 cases have been reported to health authorities, although the actual number of cases may be much higher due to significant under-reporting. Preliminary data show that the epidemic is mainly due to heterosexual transmission, and that up to 30% of cases are reported by sex workers, many of whom come from Burundi, Rwanda, Uganda and Tanzania. The ongoing transmission poses a significant risk of cross-border spread and could therefore lead to a new global smallpox epidemic, this time caused by the more virulent clade I.

The study will be carried out in collaboration with the Direction Provincial de la Santé/Kamituga and the Programme National de Lutte contre le Monkeypox et les Fièvres Virales Hémorragiques (PNLMPX/FVH) in the Kamituga Health Zone. Participants will be recruited at the Kamituga general referral hospital (HGR) or at health centers that provide mpox screening and treatment.

The MBOTE (Monkeypox Biology, Outcome, Transmission and Epidemiology) project is a multidisciplinary research collaboration between the National Institute for Biomedical Research (INRB), the Antwerp Institute of Tropical Medicine (ITM Antwerp) and the University of Antwerp.

This research protocol aims to better understand the mpox epidemic currently raging in the Kamituga SZ, as well as to provide more general information on the disease. The protocol describes the research activities that will be integrated into the ongoing epidemic investigation and control activities. Research activities will be aligned as far as possible with the ongoing epidemic response and should not hinder the response, but rather support it.

Similarly, sample collection will be aligned with the sampling carried out by the national program, and some samples will undergo additional analysis to answer the research objectives and questions.

Participation in this epidemic investigation protocol will in no way prevent patients from taking part in any other research study.

The study will be aligned as far as possible with the investigation and management of the epidemic by the national program. The study will therefore run for up to 2 months after the end of the epidemic (for convalescent patients who can be followed up for up to 2 months (day 59) after confirmation of infection), or could run for 2 years whether or not the epidemic is over. The shorter duration will be chosen, so as not to delay the reporting of results to the competent authorities, which will be essential for informing control and research activities in subsequent epidemics.

There is no fixed sample size defined for this protocol. On the contrary, as far as possible, all patients with suspected mpox will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* To be tested for VMPX at the HGR or another testing center. Patients of all ages and sexes
* Minors (≤ 17 years) are excluded from genital, anal and semen sampling and follow-up blood sampling.

Patient or culturally acceptable representative is willing and able to give informed consent for study participation.

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All persons applying to be tested for VMPX at HGR or another test center.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Characterize the clinical presentation of suspected mpox cases | Up to 2 months after the end of the epidemic, with a maximum of 2 years
  Viral Shedding Sites and Sampling Strategy: Identification of appropriate sites for viral shedding, presented as the number and types of body sites where viral shedding is detected. (qualitative measure)
  Proportion of Patients with VMPX-PCR Positivity by Sample Type: Proportion (%) of patients with VMPX-PCR positivity in each sample type (Skin swab, oropharyngeal swab, saliva, urine, semen, breast milk, anal swab, vaginal swab).
  MPXV-PCR Ct Values in Different Samples: Description of the cycle threshold (Ct) values in different types of samples. Since Ct values are numerical and specific to each sample type, you would present the Ct values for each type of sample separately.
  Duration of MPXV-PCR Positivity in Different Samples: Duration (in days) of MPXV-PCR positivity in each sample type
Characterize the longitudinal clinical course of PCR-confirmed cases | Up to 2 months after the end of the epidemic, with a maximum of 2 years
  * Frequency and Types of Complications: Measured as the percentage of patients experiencing complications (complications reported as counts or percentages).
  * In-hospital Mortality Rate and Cause of Death: Measured as the number of deaths per 100 patients, along with primary causes.
  * Duration of Signs and Symptoms: Measured in number of days from onset to resolution (could be overall or by category).
  * Frequency of Clinical Sequelae at Discharge (Day 28/59): Measured as the percentage of patients with complications at hospital discharge, Day 28, and Day 59.
  All these together will allow us to caracterise the clinical course of confirmed cases
Identification of viral shedding sites and appropriate sampling strategy | Up to 2 months after the end of the epidemic, with a maximum of 2 years
  Proportion of patients with VMPX-PCR positivity in the following samples: skin swab, oropharyngeal swab, saliva, urine, semen, breast milk, anal swab, vaginal swab Description of MPXV-PCR Ct values in different samples Duration of MPXV-PCR positivity in different samples
Characterize the virological evolution of confirmed cases | Up to 2 months after the end of the epidemic, with a maximum of 2 years
  Duration of MPXV-PCR positivity in different samples since date of diagnosis and since date of onset of symptoms Time course of CT values by sample type
Determine the seroconversion rate among confirmed cases of mpox | Up to 2 months after the end of the epidemic, with a maximum of 2 years
  Description of anti-VMPX antibody titres on days 0, 7, 14, 29 and 59 among VMPX-PCR-positive cases
Assess risk factors for mpox disease. | Up to 2 months after the end of the epidemic, with a maximum of 2 years
  Odds Ratios for Mode of Exposure: different types of exposure to mpox cases or animal reservoirs, with odds ratios calculated separately for each type of exposure.
  Odds Ratios for Socio-Demographic Factors: Odds ratios for the association between socio-demographic factors (such as age, gender, occupation) and the likelihood of mpox positivity.
  Odds Ratios for Comorbidities: odds ratios of various comorbidities (such as HIV, diabetes, etc.) and their association with mpox positivity.
  All together, these will allow us to estimate more clearly the mpox risk factors
To assess the protective effect of previous smallpox vaccination on symptomatic mpox disease. | Up to 2 months after the end of the epidemic, with a maximum of 2 years
  Vaccine efficacy based on determination of the odds ratio of vaccine status between mpox suspects tested positive and those tested negative in a test-negative case-control study.

SECONDARY OUTCOMES:
Assess genomic differences between VMPX strains isolated from confirmed cases of mpox due to sexual transmission and other modes of transmission | Up to 2 months after the end of the epidemic, with a maximum of 2 years
  Whole genome sequencing of VMPX strains from confirmed cases of mpox due to sexual transmission and other modes of transmission
Support General Referral Hospital (GRH) Kamituga | Up to 2 months after the end of the epidemic, with a maximum of 2 years
  Number of suspected and confirmed mpox cases managed at GRH Kamituga, with outcomes recorded as successful management or complications.
  Number of patients tested using the GeneXpert system, with diagnostic accuracy and turnaround time measured.
  Number of healthcare workers trained on mpox diagnosis and management, with training effectiveness assessed through pre- and post-training evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Laurens Liesenborghs, Study Director — Institute of Tropical Medicine
Locations (1):
- Kamituga General Hospital, Kamituga, Democratic Republic of the Congo

REFERENCES:
- [Background] Vakaniaki EH, Kacita C, Kinganda-Lusamaki E, O'Toole A, Wawina-Bokalanga T, Mukadi-Bamuleka D, Amuri-Aziza A, Malyamungu-Bubala N, Mweshi-Kumbana F, Mutimbwa-Mambo L, Belesi-Siangoli F, Mujula Y, Parker E, Muswamba-Kayembe PC, Nundu SS, Lushima RS, Makangara-Cigolo JC, Mulopo-Mukanya N, Pukuta-Simbu E, Akil-Bandali P, Kavunga H, Abdramane O, Brosius I, Bangwen E, Vercauteren K, Sam-Agudu NA, Mills EJ, Tshiani-Mbaya O, Hoff NA, Rimoin AW, Hensley LE, Kindrachuk J, Baxter C, de Oliveira T, Ayouba A, Peeters M, Delaporte E, Ahuka-Mundeke S, Mohr EL, Sullivan NJ, Muyembe-Tamfum JJ, Nachega JB, Rambaut A, Liesenborghs L, Mbala-Kingebeni P. Sustained human outbreak of a new MPXV clade I lineage in eastern Democratic Republic of the Congo. Nat Med. 2024 Oct;30(10):2791-2795. doi: 10.1038/s41591-024-03130-3. Epub 2024 Jun 13. PMID 38871006